CLINICAL TRIAL: NCT02233751
Title: An Open-Label Study to Evaluate the Pharmacokinetics of Testosterone Enanthate After Single-Dose Injection Via QuickShot® Testosterone in Healthy Male Subjects
Brief Title: Pharmacokinetic Study of Subcutaneous Testosterone Enanthate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Antares Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QST-14-004
Record Dates: First submitted 2014-09-02; First posted 2014-09-08 (Estimated); Results first posted 2019-04-19 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-01

CONDITIONS: Hypogonadism
Keywords: Healthy Adult Males
MeSH Terms: conditions — Hypogonadism

STUDY DESIGN:
Masking Description: The dose assignment was random among the enrolled participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Testosterone enanthate auto-injector - 50 mg (Experimental): Testosterone enanthate auto-injector - 50 mg (SC injection)
  Interventions: Combination Product: Testosterone enanthate auto-injector
- Testosterone enanthate auto-injector - 200 mg (Experimental): Testosterone enanthate auto-injector- 200 mg (SC injection)
  Interventions: Combination Product: Testosterone enanthate auto-injector

INTERVENTIONS:
Combination Product: Testosterone enanthate auto-injector — Randomization then administration of combination product study medication according to group assignment

SUMMARY:
Evaluation of pharmacokinetics of subcutaneous testosterone enanthate

DETAILED DESCRIPTION:
Evaluation of pharmacokinetics and safety profile of testosterone enanthate injected subcutaneously via auto-injector in healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male subjects, 18-55 years of age, inclusive, at the time of signing the informed consent;
* Body weight ≥50 kg and body mass index within the range 19-30 kg/m2, inclusive, at screening;
* Medically healthy subjects with clinically insignificant screening and check-in results (medical history, 12-lead electrocardiogram [ECG], physical examination, and laboratory tests); and
* Subjects who are able to understand and are willing and able to give their signed informed consent before any trial-related procedures are performed.

Exclusion Criteria:

* Currently diagnosed or a history of asthma, urticarial, angioedema, anaphylaxis, atopic dermatitis, clinically significant abnormality of skin of the abdomen, cancer, diabetes, or any other clinically significant cardiovascular, respiratory, metabolic, renal, hepatic, gastrointestinal, hematological, dermatological, venereal, neurological, psychiatric, or other major disorders;
* History of benign prostate hypertrophy (BPH), prostate cancer, or abnormal prostate specific antigen (PSA) values;
* PSA level > 3 ng/ml at screening;
* Presence or history of gastrointestinal, hepatic or renal disease, or any other condition (including surgery) known to interfere with the absorption, distribution, metabolism, or excretion of medicines;
* Systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 40 to 90 mmHg, and/or pulse rate outside the range of 40 to 100 beats per minute after one repeat at screening or check-in;
* Abnormal ECG at screening as judged by the Investigator;
* History of clinically significant drug and/or food allergies as determined by the Investigator;
* Allergy to sesame, sesame oil, or a history of hypersensitivity or idiosyncratic reaction to compounds related to the study drug
* Subjects undergoing current treatment with other androgens (i.e. dehydroepiandrosterone [DHEA]), anabolic steroids, other sex hormones, or drugs that interfere with the metabolism of testosterone (i.e. opioids, anastrozole, clomiphene, dutasteride, finasteride, flutamide, ketoconazole, spironolactone, and testolactone);
* Subjects treated within the past 12 months with estrogens, gonadotropin releasing hormone (GnRH) agonists, or growth hormone;
* Prescription, over the counter medications, vitamins, herbal and dietary supplements taken within 7 days or 5 half-lives (whichever is longer) prior to the dose of study medication and duration of the study;
* Positive screen for human immunodeficiency virus (HIV), hepatitis B, and/or hepatitis C at screening;
* Positive urine screen for drugs of abuse (amphetamine, barbiturates, benzodiazepines, cocaine, marijuana, methadone, methamphetamines, oxycodone, and opiates) or positive breath alcohol test at screening and check-in

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male
Enrollment: 12 (Actual)
Dates: Start 2014-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Jaffe, MD, Study Director — Antares Pharma Inc.
Locations (1):
- Medpace Clinical Pharmacology Unit, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pharmacokinetics of single doses of Testosterone Enanthate administered via a drug-auto injector combination product in Healthy Male Subjects
Pre-assignment Details: Two dose groups, Testosterone Enanthate 50 mg and Testosterone Enanthate 200 mg , were evaluated in parallel with 6 subjects in each dose group.
Groups:
- Testosterone Enanthate 50 mg: Testosterone enanthate auto-injector
  * 50 mg SC injection
- Testosterone Enanthate 200 mg: Testosterone enanthate auto-injector
  * 200 mg SC injection
Period: Overall Study
Arm/Group | Testosterone Enanthate 50 mg | Testosterone Enanthate 200 mg
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: In total, 12 subjects were administered study drug: 6 subjects received 50 mg SC QST and 6 subjects received 200 mg SC QST. There were no discontinuations in the study.
Groups:
- Testosterone Enanthate 50 mg: Testosterone enanthate auto-injector 50 mg
- Testosterone Enanthate 200 mg: Testosterone enanthate auto-injector 200 mg
- Total: Total of all reporting groups
Arm/Group | Testosterone Enanthate 50 mg | Testosterone Enanthate 200 mg | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.0 (11.54) | 37.5 (10.84) | 37.8 (10.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 6 | 12
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Maximum Concentration (Cmax) for Serum Testosterone and Testosterone Enanthate
Description: Cmax = Maximum blood concentration (ng/dL) of TT=Total Testosterone and TE=Testosterone Enanthate
Time Frame: Maximum serum concentrations occurring during an 8 days study window
Population: Healthy normal male volunteers
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Testosterone Enanthate 50 mg | Testosterone Enanthate 200 mg
Number analyzed (Participants) | 6 | 6
ng/dL
  Serum testosterone | 773.7 (121.26) | 1487.0 (405.34)
  Serum testosterone enanthate | 49.25 (6.90) | 267.33 (75.77)

2. Primary Outcome: Area Under the Concentration-time Curve From Time Zero to Time t
Description: AUC(0-168h) (ng⋅hr/dL) = area under the concentration-time curve from time zero to Day 8 (1 week);
Time Frame: 168 hrs
Measure: Mean (Standard Deviation); unit: (ng⋅hr/dL)
Arm/Group | Testosterone Enanthate 50 mg | Testosterone Enanthate 200 mg
Number analyzed (Participants) | 6 | 6
(ng⋅hr/dL)
  TT | 103731.5 (12591.81) | 176112.8 (47349.64)
  TE | 6122.2 (929.12) | 33535.5 (9977.18)

3. Primary Outcome: Area Under the Concentration-time Curve From Time Zero to Infinity
Description: AUC(0-inf) (ng⋅hr/dL) = area under the concentration-time curve from time zero to infinity
Time Frame: time zero to infinity
Measure: Mean (Standard Deviation); unit: (ng⋅hr/dL)
Arm/Group | Testosterone Enanthate 50 mg | Testosterone Enanthate 200 mg
Number analyzed (Participants) | 2 | 3
(ng⋅hr/dL)
  TT | 279062.2 (35973.32) | 362627.4 (138773.09)
  TE | NA (NA) — AUC(0-inf) is not calculated when the constant lambda z is not assigned, which occurs if the terminal elimination phase is not linear, if the tmax is one of the 3 last data points, or if the regression coefficient is <0.8. | 62497.5 (24618.09)

4. Secondary Outcome: Time to Maximum Concentration (Tmax)(hr)
Description: tmax = Time to reach maximum concentration
Time Frame: The sample time of Cmax during a 168 hour sampling interval
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Testosterone Enanthate 50 mg | Testosterone Enanthate 200 mg
Number analyzed (Participants) | 6 | 6
hours
  TT | 40.51 (52.95) | 19.00 (7.75)
  TE | 82.01 (53.88) | 74.00 (57.01)

5. Secondary Outcome: Half-life (t 1/2)(hr)
Description: t 1/2 = Half-life is the time required for a concentration to reduce to half its initial value
Time Frame: 168 hours
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Testosterone Enanthate 50 mg | Testosterone Enanthate 200 mg
Number analyzed (Participants) | 6 | 6
hours
  TT | 261.73 (99.04) | 131.75 (28.05)
  TE | NA (NA) — Half-life (t 1/2) is not calculated when the constant lambda z is not assigned, which occurs if the terminal elimination phase is not linear, if the tmax is one of the 3 last data points, or if the regression coefficient is <0.8. | 133.00 (67.85)

6. Secondary Outcome: Clearance CL/F (L/hr)
Description: Clearance - volume of plasma from which TT/TE is completely removed per unit time
Time Frame: 168 hours
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Testosterone Enanthate 50 mg | Testosterone Enanthate 200 mg
Number analyzed (Participants) | 6 | 6
L/hr
  TT | 18.07 (2.33) | 60.46 (21.21)
  TE | NA (NA) — Clearance - CL/F is not calculated when the constant lambda z is not assigned, which occurs if the terminal elimination phase is not linear, if the tmax is one of the 3 last data points, or if the regression coefficient is <0.8. | 352.84 (127.58)

7. Secondary Outcome: Vd/F (L)
Description: Vd/F (L) = Apparent volume of distribution
Time Frame: 168 hours
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Testosterone Enanthate 50 mg | Testosterone Enanthate 200 mg
Number analyzed (Participants) | 6 | 6
Liters
  TT | 6655.8 (1702.04) | 10959.5 (2040.99)
  TE | NA (NA) — Vd/F is not calculated when the constant lambda z is not assigned, which occurs if the terminal elimination phase is not linear, if the tmax is one of the 3 last data points, or if the regression coefficient is <0.8. | 62366.4 (23950.96)

ADVERSE EVENTS:
Time Frame: 14 days
Description: Safety assessments included adverse events and injection site assessments.
Groups:
- Treatment A: Testosterone enanthate auto-injector (SC injection) Treatment A
- Treatment B: Testosterone enanthate auto-injector (SC injections) Treatment B
Arm/Group | Treatment A | Treatment B
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 2/6 | 1/6
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A (N=6) | Treatment B (N=6)
Injection site pain (General disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other